CLINICAL TRIAL: NCT02358993
Title: The Efficacy and Cost-effectiveness of a 24-hour Course of metheNamine Hippurate for Preventing Post-Operative Urinary Tract Infection
Brief Title: Short-course Methenamine Hippurate for Prevention of Post-operative UTI
Acronym: NO-UTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 820117
Record Dates: First submitted 2015-02-03; First posted 2015-02-09 (Estimated); Results first posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Urinary Tract Infections; Catheter-Related Infections
Keywords: Urinary Tract Infections; Catheter-Related Infections; Pelvic Reconstructive Surgery; Urogynecology; Urinary catheterization; Post-operative Infections; Methenamine hippurate
MeSH Terms: conditions — Urinary Tract Infections; Catheter-Related Infections | interventions — methenamine hippurate; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methenamine (Experimental): Methenamine hippurate is a medication that exhibits antibacterial activity by converting to formaldehyde in the presence of acidic urine. It is currently FDA approved for the prophylaxis of recurrent urinary tract infections. It has been previously used in studies for prevention of UTI after gynecologic surgery. Dosage will be methenamine hippurate 1g, 1 tablet by mouth every 12 hours for 24 hours (total of two doses), with the first dose taken at least one hour prior to catheter removal.
  Interventions: Drug: methenamine hippurate
- Ciprofloxacin (Active Comparator): Ciprofloxacin is a commonly used antibiotic commonly used for prevention of UTI after catheterization. It belongs to a class of antibiotics known as the fluoroquinolones. Dosage will be ciprofloxacin 500 mg, 1 tablet by mouth every 12 hours for 24 hours (total of two doses), with the first dose taken at least one hour prior to catheter removal.
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: methenamine hippurate — A urinary antiseptic used for prevention of UTI
  Other Names: Hiprex
  Arms: Methenamine
Drug: Ciprofloxacin — An antibiotic used for treatment and prevention of UTI
  Other Names: Cipro
  Arms: Ciprofloxacin

SUMMARY:
The investigators will determine the efficacy of an innovative short regimen of methenamine hippurate on prevention of post-operative UTI in patients requiring short-term catheterization after pelvic reconstructive surgery through a single-blind, randomized controlled trial. Primary outcome will be the rate of symptomatic UTI within 3 weeks of catheter removal. The investigators will study cost-effectiveness, antibiotic resistance profiles, and adverse drug effects. Findings may reduce antibiotic use and nosocomial UTIs.

DETAILED DESCRIPTION:
Prevention of post-operative urinary tract infections (UTI) is becoming important for both the individual patient and the health system. Complications of UTI include pyelonephritis and bacteremia, requiring hospitalization and parenteral antibiotics. Additionally, recurrent exposure to antibiotics commonly given for UTIs increases the risk of antibiotic resistance to uropathogens. UTIs also increase economic burdens on the health care system, with each episode costing nearly 600 dollars. UTIs associated with catheterization are particularly costly for hospitals, resulting in decreased hospital quality measures and lack of compensation.

This is particularly important after pelvic reconstructive surgery, as reported rates of UTI reach up to 20-25%. Urinary retention requiring short-term indwelling catheterization, common in these women, contributes to the risk of UTIs by increasing the risk of bacteriuria by 5-10% per day and through the dislodging of bacterial colonies during catheter removal. Balancing prevention and resistance and cost is key. A meta-analysis by Marschall et al indicated the benefit of a short dose of antibiotic prophylaxis at catheter removal in general post-surgical patients. However, data is lacking on the effects of daily antibiotic prophylaxis on resistance and cost.

A possible alternative to antibiotics presents itself in methenamine hippurate, a urinary antiseptic which forms formaldehyde in the presence of acidic urine. It is relatively inexpensive, and does not induce resistance in vivo. Prior studies have shown that daily use of methenamine can decrease the risk of post-operative UTI.

The purpose of our study was to investigate the efficacy of a short course of methenamine hippurate at catheter removal to that of a short course of ciprofloxacin in prevention of UTIs after short-term indwelling catheterization. Additionally, we investigated factors that influence post-operative UTIs, the rate of culture-proven UTIs after prophylaxis, the antibiotic resistance profile of those undergoing prophylaxis, and the cost effectiveness of prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* female;
* patients who are able to read and write English;
* 18 years of age or older;
* underwent surgery for pelvic organ prolapse, urinary incontinence, or both;
* require post-operative short-term transurethral catheterization for greater than 24 hours.

Exclusion Criteria:

* patients undergoing surgical intervention for sacral neuromodulation, or mesh excision;
* patients requiring long-term catheterization secondary to injury to the urinary tract;
* patients who pass their post-operative trial void and thus, do not require additional catheterization;
* patients requiring catheterization for less than 24 hours;
* pregnant patients;
* patients who are breast-feeding;
* allergy to methenamine hippurate or fluroquinolones (either ciprofloxacin or levofloxacin);
* impaired renal or hepatic function;
* pre-operative urinary retention;
* patients who are currently using sulfonamides;
* patients who have severe dehydration;
* patients using tizanidine;
* patients sensitive to quinolones class;
* patients using theophylline; patients with myasthenia gravis;
* patients with prolongation of QT interval.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Chu, MD, Principal Investigator — University of Pennsylvania; Lily Arya, MD, MS, Study Director — University of Pennsylvania; Daniel Lee, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Chestnut Hill Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schiotz HA. Comparison of 1 and 3 days' transurethral Foley catheterization after retropubic incontinence surgery. Int Urogynecol J Pelvic Floor Dysfunct. 1996;7(2):98-101. doi: 10.1007/BF01902381. PMID 8798095
- [Background] Schiotz HA, Guttu K. Value of urinary prophylaxis with methenamine in gynecologic surgery. Acta Obstet Gynecol Scand. 2002 Aug;81(8):743-6. doi: 10.1080/j.1600-0412.2002.810810.x. PMID 12174159
- [Background] Anger JT, Litwin MS, Wang Q, Pashos CL, Rodriguez LV. Complications of sling surgery among female Medicare beneficiaries. Obstet Gynecol. 2007 Mar;109(3):707-14. doi: 10.1097/01.AOG.0000255975.24668.f2. PMID 17329524
- [Background] Hakvoort RA, Elberink R, Vollebregt A, Ploeg T, Emanuel MH. How long should urinary bladder catheterisation be continued after vaginal prolapse surgery? A randomised controlled trial comparing short term versus long term catheterisation after vaginal prolapse surgery. BJOG. 2004 Aug;111(8):828-30. doi: 10.1111/j.1471-0528.2004.00181.x. PMID 15270931
- [Background] Harding GK, Nicolle LE, Ronald AR, Preiksaitis JK, Forward KR, Low DE, Cheang M. How long should catheter-acquired urinary tract infection in women be treated? A randomized controlled study. Ann Intern Med. 1991 May 1;114(9):713-9. doi: 10.7326/0003-4819-114-9-713. PMID 2012351
- [Background] Saint S. Clinical and economic consequences of nosocomial catheter-related bacteriuria. Am J Infect Control. 2000 Feb;28(1):68-75. doi: 10.1016/s0196-6553(00)90015-4. PMID 10679141
- [Background] Warren JW. Catheter-associated urinary tract infections. Infect Dis Clin North Am. 1987 Dec;1(4):823-54. PMID 3333661
- [Background] Wazait HD, van der Meullen J, Patel HR, Brown CT, Gadgil S, Miller RA, Kelsey MC, Emberton M. Antibiotics on urethral catheter withdrawal: a hit and miss affair. J Hosp Infect. 2004 Dec;58(4):297-302. doi: 10.1016/j.jhin.2004.06.012. PMID 15564006
- [Background] Wolf JS Jr, Bennett CJ, Dmochowski RR, Hollenbeck BK, Pearle MS, Schaeffer AJ; Urologic Surgery Antimicrobial Prophylaxis Best Practice Policy Panel. Best practice policy statement on urologic surgery antimicrobial prophylaxis. J Urol. 2008 Apr;179(4):1379-90. doi: 10.1016/j.juro.2008.01.068. Epub 2008 Feb 20. PMID 18280509
- [Background] ACOG practice bulletin No. 104: antibiotic prophylaxis for gynecologic procedures. Obstet Gynecol. 2009 May;113(5):1180-1189. doi: 10.1097/AOG.0b013e3181a6d011. No abstract available. PMID 19384149
- [Background] Ghezzi F, Serati M, Cromi A, Uccella S, Salvatore S, Bolis P. Prophylactic single-dose prulifloxacin for catheter-associated urinary tract infection after tension-free vaginal tape procedure. Int Urogynecol J Pelvic Floor Dysfunct. 2007 Jul;18(7):753-7. doi: 10.1007/s00192-006-0233-4. Epub 2006 Nov 21. PMID 17120175
- [Background] Rogers RG, Kammerer-Doak D, Olsen A, Thompson PK, Walters MD, Lukacz ES, Qualls C. A randomized, double-blind, placebo-controlled comparison of the effect of nitrofurantoin monohydrate macrocrystals on the development of urinary tract infections after surgery for pelvic organ prolapse and/or stress urinary incontinence with suprapubic catheterization. Am J Obstet Gynecol. 2004 Jul;191(1):182-7. doi: 10.1016/j.ajog.2004.03.088. PMID 15295362
- [Background] Baertschi U, Kunz J. [Comparative study on the question of systemic chemoprophylaxis following gynecological surgery]. Schweiz Med Wochenschr. 1976 Mar 13;106(11):380-5. German. PMID 1251156
- [Background] Gordon KA, Jones RN; SENTRY Participant Groups (Europe, Latin America, North America). Susceptibility patterns of orally administered antimicrobials among urinary tract infection pathogens from hospitalized patients in North America: comparison report to Europe and Latin America. Results from the SENTRY Antimicrobial Surveillance Program (2000). Diagn Microbiol Infect Dis. 2003 Apr;45(4):295-301. doi: 10.1016/s0732-8893(02)00467-4. PMID 12730002
- [Background] Tyreman NO, Andersson PO, Kroon L, Orstam S. Urinary tract infection after vaginal surgery. Effect of prophylactic treatment with methenamine hippurate. Acta Obstet Gynecol Scand. 1986;65(7):731-3. doi: 10.3109/00016348609161491. PMID 3544661
- [Background] Knoff T. [Methenamine hippurate. Short-term catheterization in gynecologic surgery. A double-blind comparison of Hiprex and placebo]. Tidsskr Nor Laegeforen. 1985 Mar 10;105(7):498-9. No abstract available. Norwegian. PMID 3887639
- [Background] Ladehoff P, Jacobsen JC, Olsen H, Pedersen GT, Sorensen T. [The preventive effect of methenamine hippurate (Haiprex) on urinary infections after short-term catheterization. A clinical study]. Ugeskr Laeger. 1984 May 7;146(19):1433-4. No abstract available. Danish. PMID 6515752
- [Background] Strom JG Jr, Jun HW. Effect of urine pH and ascorbic acid on the rate of conversion of methenamine to formaldehyde. Biopharm Drug Dispos. 1993 Jan;14(1):61-9. doi: 10.1002/bdd.2510140106. PMID 8427945
- [Background] Marschall J, Carpenter CR, Fowler S, Trautner BW; CDC Prevention Epicenters Program. Antibiotic prophylaxis for urinary tract infections after removal of urinary catheter: meta-analysis. BMJ. 2013 Jun 11;346:f3147. doi: 10.1136/bmj.f3147. PMID 23757735
- [Background] Sutkin G, Alperin M, Meyn L, Wiesenfeld HC, Ellison R, Zyczynski HM. Symptomatic urinary tract infections after surgery for prolapse and/or incontinence. Int Urogynecol J. 2010 Aug;21(8):955-61. doi: 10.1007/s00192-010-1137-x. Epub 2010 Mar 31. PMID 20354678
- [Background] Dieter AA, Amundsen CL, Edenfield AL, Kawasaki A, Levin PJ, Visco AG, Siddiqui NY. Oral antibiotics to prevent postoperative urinary tract infection: a randomized controlled trial. Obstet Gynecol. 2014 Jan;123(1):96-103. doi: 10.1097/AOG.0000000000000024. PMID 24463669
- [Background] Turck M, Stamm W. Nosocomial infection of the urinary tract. Am J Med. 1981 Mar;70(3):651-4. doi: 10.1016/0002-9343(81)90590-8. PMID 7011018
- [Background] Duclos JM, Larrouturou P, Sarkis P. Timing of antibiotic prophylaxis with cefotaxime for prostatic resection: better in the operative period or at urethral catheter removal? Am J Surg. 1992 Oct;164(4A Suppl):21S-23S. doi: 10.1016/s0002-9610(06)80053-x. PMID 1443356
- [Background] Lusardi G, Lipp A, Shaw C. Antibiotic prophylaxis for short-term catheter bladder drainage in adults. Cochrane Database Syst Rev. 2013 Jul 3;2013(7):CD005428. doi: 10.1002/14651858.CD005428.pub2. PMID 23824735
- [Background] Lee BS, Bhuta T, Simpson JM, Craig JC. Methenamine hippurate for preventing urinary tract infections. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD003265. doi: 10.1002/14651858.CD003265.pub3. PMID 23076896
- See also: Methenamine. In: Lexi-Drugs Online. Hudson, OH: Lexi-Comp, Inc. [updated 2/1/14; accessed 2/21/14]. — http://online.lexi.com/lco/action/doc/retrieve/docid/patch_f/7265?hl=6550/
- See also: Methenamine. In: Micromedex 2.0. Martindale - The Complete Drug Reference. Ann Arbor, MI: Truven Health Analytics. [updated 8/20/2010; accessed 2/21/14]. — http://www.micromedexsolutions.com/micromedex2/librarian/
- See also: Nitrofurantoin. In: Micromedex 2.0. Martindale - The Complete Drug Reference. Ann Arbor, MI: Truven Health Analytics. [updated 8/20/2010; accessed 2/21/14]. — http://www.micromedexsolutions.com/micromedex2/librarian/
- See also: Ciprofloxacin. In: Micromedex 2.0. Martindale - The Complete Drug Reference. Ann Arbor, MI: Truven Health Analytics. [updated 8/20/2010; accessed 2/21/14]. — http://www.micromedexsolutions.com/micromedex2/librarian/
- See also: Sulfamethoxazole/Trimethoprim. In: Micromedex 2.0. Martindale - The Complete Drug Reference. Ann Arbor, MI: Truven Health Analytics. [updated 8/20/2010; accessed 2/21/14]. — http://www.micromedexsolutions.com/micromedex2/librarian/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methenamine | Ciprofloxacin
Started | 105 | 96
Completed | 103 | 94
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methenamine | Ciprofloxacin | Total
Number analyzed (Participants) | 103 | 94 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: In the Ciprofloxacin group, one age datapoint was missing from the dataset.
  years
    number analyzed (Participants) | 103 | 93 | 196
    (all) | 63.9 (10.7) | 61.6 (10.5) | 62.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 94 | 197
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Missing race data on 1 participant randomized to the Ciprofloxin arm and 2 participants randomized to the methenamine hippurate arm.
  Participants
    number analyzed (Participants) | 101 | 93 | 194
    Caucasion | 83 | 72 | 155
    Black | 15 | 18 | 33
    Asian American/Pacific Islander | 2 | 1 | 3
    Did not answer | 1 | 2 | 3
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (4.9) | 28 (5.3) | 27.6 (5.1)
Postmenopausal [Count of Participants; unit: Participants] | 83 | 71 | 154
Current Smoker [Count of Participants; unit: Participants] | 3 | 5 | 8
History of recurrent UTI [Count of Participants; unit: Participants] | 4 | 4 | 8
Recent preoperative UTI [Count of Participants; unit: Participants] | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Treatment of Clinically Suspected UTI - Using Intent to Treat Analysis
Description: This is defined as any symptomatic UTI requiring treatment with antibiotics as determined by the development of 2 or more of the following symptoms, in the absence of vaginal symptoms: urinary frequency; urinary urgency; dysuria; fever over 38oC/100.4oF; suprapubic, flank, or back pain; and/or chills.
Time Frame: 3 weeks post-operative
Population: Intent to Treat model
Measure: Count of Participants; unit: Participants
Arm/Group | Methenamine | Ciprofloxacin
Number analyzed (Participants) | 101 | 93
Participants | 13 | 12
Statistical Analysis 1: Comparison: Methenamine vs Ciprofloxacin; Test type: Non-Inferiority — Non-inferiority of the primary outcome was achieved if the lower limit of the 95% confidence interval of the mean difference was greater than the specified non-inferiority margin of 15%(a clinically relevant margin within the range of those commonly used in non-inferiority and equivalence trials for studies examining antibiotic use for UTI); Risk Ratio (RR) = -.01

2. Primary Outcome: Treatment of Clinically Suspected UTI - Per Protocol
Description: as for outcome 1
Time Frame: 3 weeks post-operative
Population: Per protocol model
Measure: Count of Participants; unit: Participants
Arm/Group | Methenamine | Ciprofloxacin
Number analyzed (Participants) | 98 | 89
Participants | 12 | 12

3. Secondary Outcome: Number of Participants With Culture-positive Symptomatic UTI
Description: All patients will be encouraged to submit urine cultures prior to treatment, but this is not always possible. Amongst patients who undergo urine culture as part of standard of care for UTI, the rate of positive cultures will be identified.
Time Frame: 3 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Methenamine | Ciprofloxacin
Number analyzed (Participants) | 101 | 93
Participants | 5 | 4

4. Secondary Outcome: Antibiotic Resistance of Culture-positive Symptomatic UTI
Description: All patients who submit urine cultures that are positive will have sensitivities performed as per standard care. The prevalence of bacterial species and sensitivities will be collected
Time Frame: 3 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Methenamine | Ciprofloxacin
Number analyzed (Participants) | 101 | 93
Participants | 0 | 0

5. Secondary Outcome: Cost-effectiveness of Prophylaxis With Methenamine Hippurate for Prevention of Post-operative UTI Compared to Prophylaxis With Fluoroquinolones
Description: Routine costs of prevention of UTI with methenamine hippurate prophylaxis will be compared with costs of prevention of UTI with fluoroquinolone prophylaxis. We plan to capture costs for each direct medical service use, direct non-medical items, and indirect items related to post-operative UTIs in each arm of the trial.
Time Frame: 3 weeks post-operative
Population: The data for this secondary was not collected. No costs were captured.
Arm/Group | Methenamine | Ciprofloxacin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Prevalence of Side Effects
Description: Adverse effects from the administration of methenamine and fluoroquinolones will be collected.
Time Frame: within 24 hours of administration
Population: The data for this secondary outcome measure was not collected.
Arm/Group | Methenamine | Ciprofloxacin
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Rate of UTI Consistent With NHSN Criteria
Description: We plan to analyze the prevalence of UTI in this population that meet the definitions of symptomatic UTI and catheter-associated UTI according to the National Healthcare Safety Network criteria.
Time Frame: 3 weeks post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Methenamine | Ciprofloxacin
Number analyzed (Participants) | 101 | 93
Participants | 10 | 6

ADVERSE EVENTS:
Time Frame: The AEs were collected from time of surgery to their clinical post-operative visit, usually between 4 and 12 weeks post-op.
Arm/Group | Methenamine | Ciprofloxacin
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/94
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/94
Other Adverse Events (participants affected / at risk) | 0/103 | 3/94
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methenamine (N=103) | Ciprofloxacin (N=94)
nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT02358993/Prot_SAP_000.pdf
  • Informed Consent Form (2017-04-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT02358993/ICF_001.pdf